CLINICAL TRIAL: NCT05927025
Title: Evaluation of Different NiTi Rotary Files With NiTi Hand Files to Postoperative Pain Effects : A Randomized Controlled Clinical Trial
Brief Title: Can the Different Instruments Used ın Root Canal Treatment Have an Effect on Postoperative Pain?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Merve Abakli Inci, assistant professor, Necmettin Erbakan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NecmettinMA-001
Record Dates: First submitted 2023-06-03; First posted 2023-07-03 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Postoperative Pain
Keywords: Root canal treatment; Nickel-Titanium instruments; Postoperative pain; Primary tooth
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant
Masking Description: Masking was applied only to the patients and their parents included in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Hand K-files (Experimental): NiTi K type hand file (Perfect Medical Instrument Co., Ltd. Shenzhen, China), Contrary to stainless steel files, turning is produced with the buckling method. torsional resistance and bending resistance of files compared to stainless steel files found more successful in comparison. 16 mm of the files are finished It has the edge. Our Work is 25mm long; 15K (white), 20K (yellow), 25K (red), 30 K (blue) files were used. NiTi K type #15, #20, #25, and #30 hand files were used with a quarter-turn pulling motion, respectively.
  Interventions: Procedure: Hand K-files
- ProTaper Next (Experimental): The ProTaper Next (PTN) system is produced by adding M-Wire alloy to the ProTaper Universal (PU) system. With the M-Wire alloy, it is aimed to increase the flexibility and cyclic fatigue resistance of the files. The combination of three important design features in PTN files, including changing taper on a single file, M-wire technology and offset design, is one of the important features that distinguish it from other files. PTN X1 and X2 files have both an ascending and a descending conical design on a single file; PTN X3, X4 and X5 files have a constant taper from D1-D3, then taper design that tapers off over the rest of their active segments.
  Interventions: Procedure: Hand K-files
- WaveOne Gold (Experimental): They are produced by applying Gold-wire process to the WaveOne (WO) system. The WOG file system exhibits repetitive back-and-forth mutual 'reciprocation' motion during preparation, in contrast to the continuous rotational motion. While rotating 150° counterclockwise during the reciprocating motion, clockwise It turns 30° in the direction of, and after 3 cycles, it completes 1 full cycle. Thus, it contributed positively to the file reaching the apical without applying excessive pressure, increasing the cutting efficiency, and accelerating the coronal movement of the debris. Small (yellow-20/0.07), WO Primary (red-25/0.07), and WOG Medium (green-35/0.06) files were used with the appropriate speed and torque values recommended by the manufacturer (300 rpm and 2.0 Ncm) by applying crown down technique. WOG files were operated in a reciprocating motion (150° counterclockwise, 30° clockwise).
  Interventions: Procedure: Hand K-files
- AF Baby Rotary File (Experimental): AF Baby rotary file is specially designed for milk teeth. Entry file 11 mm other the files are 16 mm long and consist of 4 different rotary instruments; (17/.08), (20/.04), (25/.04) and (30/.04).The cross-sections of the files are triangular and heat treatment is applied to the NiTi wire. produced as a result. Thus, an increase in resistance to cyclic fatigue and an increase in dentin It is aimed to reduce screwing. Root canal thanks to its flexibility It adapts very well to the curvatures in its anatomy. AF Baby rotary files #20, #25, and #30 were used with the crown down technique with the appropriate speed and torque values (350 rpm and 2.0 Ncm) recommended by the manufacturer.
  Interventions: Procedure: Hand K-files
- EndoArt NiTi Pedo Golf File (Experimental): EndoArt NiTi Pedo Gold file is specially designed for primary teeth. 18mm length consists of 4 different rotary tools: (15/06) white, (20/04) yellow, (25/04) red, (30/04) blue. The cross-sections of the files are triangular, and Gold wire technology is used in the production phase. were produced using Thus, a titanium oxide layer on the surface of the instrument Happened. Thus, it is more flexible and more flexible than conventional NiTi alloys. resistant and 2 times better cyclic fatigue resistance than conventional files exists. EndoArt NiTi Pedo Golf File; EndoArt NiTi Pedo Gold #15, #20, and #30 files were used with the crown down technique with the appropriate speed and torque values recommended by the manufacturer (350 rpm and 2.0 Ncm).
  Interventions: Procedure: Hand K-files

INTERVENTIONS:
Procedure: Hand K-files — It is used for cleaning and shaping root canals.
  Other Names: ProTaper Next; WaveOne Gold; AF Baby Rotary File; EndoArt NiTi Pedo Golf File

SUMMARY:
Root canal treatment is a treatment method in which the pulp is irreversibly infected due to caries or trauma or when the pulp loses its vitality. Biomechanical preparation of primary teeth is an important step for a successful root canal treatment. The success of root canal treatment depends not only on the biological results of the treatment, but also on minimizing the postoperative pain of the patients. Therefore, the elimination of factors associated with postoperative pain has an important role in the prognosis of patients after treatment. In all root canal preparation methods, some debris overflows from the apical. Debris protruding into the apical area causes postoperative pain. Many studies in the literature have shown that NiTi rotary files cause less extrusion of debris compared to hand files, and therefore less postoperative pain. Within the scope of this study, the effect of NiTi K hand file and WaveOne Gold, ProTaper Next, EndoArt NiTi Pedo Gold file, AF Baby rotary file systems on postoperative pain in root canal treatment preparations applied to the mandibular primary molar teeth of pediatric patients aged 5-8 years. It is intended to be evaluated using VAS).

In our research; ProTaper Next (PTN), WaveOne Gold (WOG), AF Baby rotary file, EndoArt NiTi Pedo Gold file, NiTi K type hand files were used. 100 patients between the ages of 5 and 8 who had root canal treatment indications for mandibular primary second molars were included in the study. The patients were divided into 5 groups with 20 patients in each group. All systems were used according to the manufacturer's instructions and all treatments were performed by a single operator in a single session. Postoperative pain was recorded using the Visual Analog Scale (VAS) at the 6th, 12th, 18th, 24th, 48th, 72nd hour and 1st week following treatment. The obtained data were evaluated statistically.

ELIGIBILITY:
Inclusion Criteria:

* No analgesic use 12 hours before root canal treatment
* No systemic disease.
* Teeth with a diagnosis of irreversible pulpitis, no other teeth causing pain at the site of the tooth to be treated, no inter-root bone loss exceeding 1/3, and root canal inclinations of no more than 25° according to Schneider method were included in the study.

Exclusion Criteria:

* Patients with post-procedural analgesic use were excluded from the study
* Patients whose parents did not fully understand the instructions and who did not attend the follow-up visit one week after treatment were excluded.

Ages: 5 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2023-01-18 (Actual)

PRIMARY OUTCOMES:
Postoperative Pain Assessments | 6 hours
  Evaluation of the effect on pain after root canal treatment; Parents were trained to use the pain scale; Postoperative pain occurring at the 6th hour was evaluated. All parents participating in the study were blinded to the treatment protocol used for the children. Evaluation of postoperative pain was performed using the VAS . It was explained that the closest score between "0" no pain and "10" severe pain scores should be recorded by the parents.
Postoperative Pain Assessments | 12 hours
  Evaluation of the effect on pain after root canal treatment; Parents were trained to use the pain scale; Postoperative pain occurring at the 12th hour was evaluated. All parents participating in the study were blinded to the treatment protocol used for the children. Evaluation of postoperative pain was performed using the VAS. It was explained that the closest score between "0" no pain and "10" severe pain scores should be recorded by the parents.
Postoperative Pain Assessments | 24 hours
  Evaluation of the effect on pain after root canal treatment; Parents were trained to use the pain scale; Postoperative pain occurring at the 24th hour was evaluated. All parents participating in the study were blinded to the treatment protocol used for the children. Evaluation of postoperative pain was performed using the VAS. It was explained that the closest score between "0" no pain and "10" severe pain scores should be recorded by the parents.
Postoperative Pain Assessments | 48 hours
  Evaluation of the effect on pain after root canal treatment; Parents were trained to use the pain scale; Postoperative pain occurring at the 48th hour was evaluated. All parents participating in the study were blinded to the treatment protocol used for the children. Evaluation of postoperative pain was performed using the VAS. It was explained that the closest score between "0" no pain and "10" severe pain scores should be recorded by the parents.
Postoperative Pain Assessments | 72 hours
  Evaluation of the effect on pain after root canal treatment; Parents were trained to use the pain scale; Postoperative pain occurring at the 72nd hour was evaluated. All parents participating in the study were blinded to the treatment protocol used for the children. Evaluation of postoperative pain was performed using the VAS. It was explained that the closest score between "0" no pain and "10" severe pain scores should be recorded by the parents.
Postoperative Pain Assessments | 1 weeks
  Evaluation of the effect on pain after root canal treatment; Parents were trained to use the pain scale; Postoperative pain occurring at the 1st week was evaluated. All parents participating in the study were blinded to the treatment protocol used for the children. Evaluation of postoperative pain was performed using the VAS. It was explained that the closest score between "0" no pain and "10" severe pain scores should be recorded by the parents.

CONTACTS AND LOCATIONS:
Locations (1):
- Necmettin Erbakan University, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The research will be published soon.